CLINICAL TRIAL: NCT02068378
Title: Clinical Evaluation of Visual Feedback With Optical Sensing in Lung Cancer Patients Undergoing Radiotherapy: A Feasibility Study
Brief Title: Visual Feedback With Optical Sensing - A Feasibility Study
Acronym: ROSS-LC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sally Falk (Other)
Responsible Party: Sponsor-Investigator, Sally Falk, Clinical Trials Project Manager, The Christie NHS Foundation Trust
Organization: The Christie NHS Foundation Trust (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 13_DOG07_158; CFTSp076 (Other: The Christie NHS Foundation Trust)
Record Dates: First submitted 2014-02-18; First posted 2014-02-21 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CMPE Optical Sensor Device (Experimental): Single arm study
  Interventions: Device: CMPE Optical Sensor Device

INTERVENTIONS:
Device: CMPE Optical Sensor Device — Christie Medical Physics & Enginieering visual feedback with optical sensing device.

SUMMARY:
Lung cancer is the second most common cancer in the United Kingdom with around 40,000 new cases diagnosed every year. Lung cancer is associated with a very poor prognosis (<10% patient survival at 5 years). New strategies are urgently needed to improve survival in this group of patients.

The most effective and common treatment for lung cancer is radiotherapy (either alone or combined with chemotherapy and/or surgery) and generally high doses of radiotherapy are given to the tumour. However, increasing the radiotherapy dose carries an increased risk of damage to the surrounding healthy tissue. Damage can be minimised by reducing movement within the lung, caused by factors such as breathing and patient motion, during treatment.

This study tests a new medical device that has been developed to monitor and help patients control their breathing and movement during treatment. Optical sensors will detect any motion of the patient's torso and this will be fed back to the patient in the form of a visual aid allowing them to regulate their breathing and maintain their ideal treatment position.

The device has already been shown to reduce motion in healthy volunteers. In this study the investigators hope to demonstrate that the visual aids are tolerable in lung cancer patients. The investigators additionally aim to show the device will help reduce movements of the chest and also the lung tumour, leading to improvements in treatment results.

DETAILED DESCRIPTION:
In this study each participant will undergo 4 imaging sessions (one training session and 3 study sessions) where participants will be asked to use the optical feedback display to regulate breathing patterns.

The training session and each study session will proceed as follows:

* The patient receives standard treatment including any pre-treatment Cone Beam CT (CBCT) imaging.
* The patient is allowed to get up off the treatment couch and relax whilst the sensor device is turned on.
* The patient is set-up again.
* The patient is asked to free-breathe (i.e. breathe normally) and the surface motion is recorded using the optical sensor. The first 30 seconds are used to generate the reference surface used throughout the rest of the process. A 4D CBCT scan is acquired during free-breathing to assess tumour motion.
* The patient is then asked to control their breathing using the feedback displays and data is recorded for ~1:30 minutes in each case.
* A 4D CBCT scan will be acquired during controlled breathing with the traffic light feedback visualization scheme to assess tumour motion.

ELIGIBILITY:
Inclusion Criteria:

* Stage 1-3 lung cancer (Non Small Cell Lung Cancer and Small Cell Lung Cancer; histological diagnosis not mandatory) including at least 5 patients with lower lobe tumours
* Suitable for radical radiotherapy
* Tumour judged inoperable by a thoracic surgeon
* At least 18 years old

Exclusion Criteria:

* Stage 4 Non Small Cell Lung Cancer
* Unable to give informed consent
* Epilepsy or migraine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-04-30 (Actual); Primary Completion 2016-02-28 (Actual); Study Completion 2016-02-28 (Actual)

PRIMARY OUTCOMES:
Tolerability of the device assessed as the percentage of patients who complete all 3 study sessions | 6 months

SECONDARY OUTCOMES:
Reduction of periodic respiratory motion body surface amplitude using the device as compared to free breathing. | 6 months
Reduction of overall body surface variability using the device as compared to free breathing. | 6 months
Reduction in internal tumour motion magnitude and variability using the device as compared to free-breathing. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gareth Price, PhD, Principal Investigator — The Christie NHS Foundation Trust
Locations (1):
- The Christie NHS Foundation Trust, Manchester, Greater Manchester, United Kingdom